CLINICAL TRIAL: NCT03952221
Title: Effects of Various Types of Ultrasound Therapy in Hip Osteoarthritis - a Double-blinded, Placebo-controlled, Follow-up Study
Brief Title: Effects of Various Types of Ultrasound Therapy in Hip Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Petz Aladar County Teaching Hospital (Other)
Responsible Party: Principal Investigator, Márta Király, chief physician, Petz Aladar County Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PetzAladarCountyTH
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Hip Osteoarthritis
Keywords: hip osteoarthritis; sonotens; pulsed ultrasound; continuous ultrasound
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual physiotherapy and continuous ultrasound therapy (Active Comparator): Patients received usual physiotherapy (exercise, massage, balneotherapy) and continuous ultrasound therapy (BTL-4825S Premium device, head size of 5 cm2, 3 MHz frequency, 1,5 W/cm2 SATA intensity) every working day for two weeks (10 occasions).
  Interventions: Device: Continuous ultrasound therapy
- Usual physiotherapy and pulsed ultrasound therapy (Active Comparator): Patients received usual physiotherapy (exercise, massage, balneotherapy) and pulsed ultrasound therapy (BTL-4825S Premium device, head size of 5 cm2, 3 MHz frequency, 1,5 W/cm2 SATA intensity, 50% duty cycle) every working day for two weeks (10 occasions).
  Interventions: Device: pulsed ultrasound therapy
- Usual physiotherapy and sonotens therapy (Active Comparator): Patients received usual physiotherapy (exercise, massage, balneotherapy) and sonotens therapy (BTL-4825S Premium device, head size of 5 cm2, 3 MHz frequency, 0,5 W/cm2 SATA intensity, transcutanous electrical nerve stimulation) every working day for two weeks (10 occasions).
  Interventions: Device: US and electrotherapy (sonotens)
- Usual physiotherapy and sham ultrasound therapy (Placebo Comparator): Patients received usual physiotherapy (exercise, massage, balneotherapy) and sham ultrasound therapy (BTL-4825S Premium device, head size of 5 cm2, 0 MHz frequency, 0 W/cm2 SATA intensity) every working day for two weeks (10 occasions).
  Interventions: Device: Sham ultrasound therapy

INTERVENTIONS:
Device: Continuous ultrasound therapy — continuous US therapy once a day, 9 minutes/session for two weeks (10 occasions) with BTL-4825S Premium device, 5 cm2 probe, 3 MHz frequency, 1,5 W/cm2 SATA intensity
  Arms: Usual physiotherapy and continuous ultrasound therapy
Device: pulsed ultrasound therapy — pulsed US therapy once a day, 9 minutes/session, for two weeks (10 occasions) with BTL-4825S Premium device, 5 cm2 probe, 3 MHz frequency, 1,5 W/cm2 SATA intensity, 50% duty cycle
  Arms: Usual physiotherapy and pulsed ultrasound therapy
Device: US and electrotherapy (sonotens) — US and electrotherapy (transcutaneous electrical nerve stimulation) once a day, 10 minutes /session, for two weeks (10 occasions) with BTL-4825S Premium device, 5 cm2 probe, US: 3 MHz frequency, 0,5 W/cm2 SATA intensity, TENS: application in conventional mode at 100 Hz frequency and 100 μs wavelength
  Arms: Usual physiotherapy and sonotens therapy
Device: Sham ultrasound therapy — sham US therapy once a day for two weeks (10 occasions) with BTL-4825S Premium device, 5 cm2 probe, 0 MHz frequency, 0 W/cm2 SATA intensity
  Arms: Usual physiotherapy and sham ultrasound therapy

SUMMARY:
This study evaluates the effects of various types of ultrasound therapy: continuous, pulsed, sham ultrasound and ultrasound combined with electrotherapy in patients with hip osteoarthritis. Beside ultrasound therapy, patients received usual physiotherapy (balneotherapy, exercise and massage) either.

DETAILED DESCRIPTION:
During ultrasound therapy electrical energy is converted into mechanical energy and heat. It has physical, chemical and biologic effects, like thermal effect, micro-massage, increased tissue metabolism, capillary permeability and tissue healing. Continuous or pulsed forms can be applied.

As pulsed ultrasound therapy has no thermal effect, greater intensity can be used. It can alleviate acute pain and inflammation. Continuous ultrasound is usually used in chronic musculoskeletal diseases, in case of limitation of joint motion because its thermal effect.

Ultrasound can be combined with electrotherapy, when the effects of the two modalities are summed up.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age with moderate hip osteoarthritis (radiologically Kellgren- Laurence II-III. stage)
* chronic hip pain (for at least 8 weeks)
* pain intensity is ≥ 50mm on a Visual Analogue Scale
* no physiotherapy or local injection (steroid, hialuronic acid) within 3 months before starting the study

Exclusion Criteria:

* acute hip pain (duration is less than 8 weeks)
* steroid, hialuronic acid injection into the hip joint within 3 months
* physiotherapy of the hip within 3 months
* inflammatory hip osteoarthritis
* infection
* fever
* tumour
* epilepsy
* pregnancy
* untreated hypertension
* heart failure (NYHA II-IV. stage)
* inflammatory rheumatic diseases
* hip arthroplasty
* pacemaker or intracardiac device
* severe osteoporosis
* osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-08-03 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
change in severity of pain at rest | Week 0 and Week 2
  change from baseline severity of pain at rest recorded on a 100 mm visual analogue scale, where 0 mm represents no pain, 100 mm represents unbearable pain.
change in severity of pain at rest | Week 0 and Week 12
  change from baseline severity of pain at rest recorded on a 100 mm visual analogue scale, where 0 mm represents no pain, 100 mm represents unbearable pain.
change in function | Week 0 and Week 2
  change from baseline Western Ontario and McMaster Universities Arthritis Index (WOMAC) at week 2. It is comprised of 24 items divided into three subscales: Pain (5 items), stiffness (2 items), and physical function (17 items). All the items are scored on a 100mm visual analogue scale. Values are summed up for a combined WOMAC score. The lower score represents better outcome.
change in function | Week 0 and Week 12
  change from baseline Western Ontario and McMaster Universities Arthritis Index (WOMAC) at week 12. It is comprised of 24 items divided into three subscales: Pain (5 items), stiffness (2 items), and physical function (17 items). All the items are scored on a 100mm visual analogue scale. Values are summed up for a combined WOMAC score. The lower score represents better outcome.
change in function | Week 0 and Week 2
  change from baseline physical function measured by the 6-minute walking test. The test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. Patients can walk at a self chosen walking speed, can have a rest or can use a walking aid. The accomplished distance is the total distance at the end of the 6 minutes.
change in function | Week 0 and Week 12
  change from baseline physical function measured by the 6-minute walking test at Week 12. The test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. Patients can walk at a self chosen walking speed, can have a rest or can use a walking aid. The accomplished distance is the total distance at the end of the 6 minutes.
change in quality of life | Week 0 and Week 2
  change from baseline quality of life (36-Item Short Form Health Survey /SF-36/) at week 2. It consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more the disability, i.e. a score of zero is equivalent to maximum disability.
change in quality of life | Week 0 and Week 12
  change from baseline quality of life (36-Item Short Form Health Survey /SF-36/) at week 12. It consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more the disability, i.e. a score of zero is equivalent to maximum disability.

CONTACTS AND LOCATIONS:
Overall Officials: Márta Király, Principal Investigator — Petz Aladar County Teaching Hospital
Locations (2):
- Hungary (2):
  - Petz Aladár County Teaching Hospital, Győr
  - Zsigmondy Vilmos Harkány Spa Hospital, Harkány